CLINICAL TRIAL: NCT00006469
Title: Phase II Trial of Concurrent Paclitaxel, Carboplatin and External Beam Radiotherapy Followed by Surgical Resection in Stage IIIA (N2) Non-small Cell Lung Cancer
Brief Title: Combination Chemotherapy and Radiation Therapy Followed By Surgery in Treating Patients With Stage IIB or Stage IIIA Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: David J. Perry, MD, Washington Cancer Institute at Washington Hospital Center
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: CDR0000068288; WHC-99444; NCI-V00-1632
Record Dates: First submitted 2000-11-06; First posted 2003-01-27 (Estimated); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Lung Cancer
Keywords: stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Concurrent Paclitaxel, Carboplatin, and External-Beam Radiation Followed by Surgical Resection in Locally Advanced Non-Small-Cell Lung Cancer
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm study (Other): Concurrent Paclitaxel, Carboplatin, and External-Beam Radiation Followed by Surgical Resection in Locally Advanced Non-Small-Cell Lung Cancer
  Interventions: Drug: carboplatin; Drug: paclitaxel; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin
  Other Names: paraplatin
Drug: paclitaxel
  Other Names: taxol
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining these treatments before surgery may kill more tumor cells in patients with non-small cell lung cancer.

PURPOSE: Phase II trial to study the effectiveness of combining chemotherapy with radiation therapy before surgery in treating patients who have stage IIB non-small cell lung cancer or stage IIIA non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate, duration of response, and survival in patients with bulky stage IIB or stage IIIA non-small cell lung cancer treated with paclitaxel, carboplatin, and radiotherapy followed by surgical resection.
* Assess the toxicity of this regimen in this patient population.

OUTLINE: This is a multicenter study.

Patients receive paclitaxel IV over 1 hour and carboplatin IV over 30 minutes weekly for 5 weeks. Patients also undergo concurrent radiotherapy daily 5 days a week for 5 weeks in the absence of unacceptable toxicity. At approximately 4 weeks after completion of chemoradiotherapy, patients with stable or regressive disease undergo surgical resection. If disease is unresectable, patients receive an additional 2 weeks of radiotherapy.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 29-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed bulky stage IIB or stage IIIA non-small cell lung cancer

  * Ipsilateral mediastinal node involvement by mediastinoscopy
* No contralateral lymph node involvement
* No malignant pleural effusion
* No distant metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* ALT/AST less than 2 times upper limit of normal
* Bilirubin no greater than 1.5 mg/dL

Renal:

* Creatinine no greater than 2.0 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other prior malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix or nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1999-08; Primary Completion 2006-01-30 (Actual); Study Completion 2006-01-30 (Actual)

PRIMARY OUTCOMES:
Pathologic response rate | 3-5 Years
  as measured by pathology of the resected specimen and chest x-ray at 3 and 5 years after completion of study treatment.
Disease-free and overall survival at 3 and 5 years after completion of study treatment | 3-5 Years

CONTACTS AND LOCATIONS:
Overall Officials: David J. Perry, MD, Study Chair — Medstar Health Research Institute
Locations (2):
- United States (2):
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Harry and Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center, Baltimore, Maryland